CLINICAL TRIAL: NCT01659372
Title: Phase 1 Study of Low Level Laser Therapy Versus Naproxen
Brief Title: Low Level Laser Therapy Versus Pharmacotherapy in in Improving Masticatory Muscle Pain
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, saranaz azari-marhabi, oral medicine resident, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABT-1233-RV
Record Dates: First submitted 2012-08-04; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: TMD
Keywords: temporomandibular disorder; myofascial pain syndrome
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myofascial Pain Syndromes | interventions — Low-Level Light Therapy; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low level laser therapy (Experimental): this arm recieves low level laser therapy treatment for 12 sessions.
  Interventions: Radiation: low level laser therapy
- naproxen (Experimental): this arm takes naproxen 500 mg twice daily for 3weeks
  Interventions: Drug: Naproxen

INTERVENTIONS:
Radiation: low level laser therapy
  Arms: Low level laser therapy
Drug: Naproxen
  Arms: naproxen

SUMMARY:
tempromandibuar disorders are a group of heterogenous pathologies affecting temporomandibular joint,muscles or both.in more than 90%of cases muscles are the origin of pain.TMDs cause pain,movement disability and deficit in quality of life.in more than 90%of cases pain is the major complaint.we run this investigation to find the analgesic effct of low level laser therapy versus pharmacotherapy with naproxen in improving pain.

ELIGIBILITY:
Inclusion Criteria:

* patients with TMD affecting masticatory muscles

Exclusion Criteria:

* systemic disease
* GI problem
* pregnancy
* epidermal cancer

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
reduction of paim measured by VAS | 1 month
  VAS is visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Beheshti University, Tehran, Iran